CLINICAL TRIAL: NCT04625686
Title: A Multi-Site, Non-Interventional Study to Compare the Outcomes of Psychiatric Treatment of Suicidal Adolescents in Different Treatment Settings
Brief Title: Observational Study to Compare Outcomes of Different Psychiatric Treatment of Suicidal Adolescents
Acronym: Pre-START
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-0686
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Results first posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-08

CONDITIONS: Suicidal Ideation
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Inpatient Treatment: Inpatient psychiatric treatment
  Interventions: Behavioral: Mental Health Treatment
- OCIC Treatment: In-person outpatient crisis intervention
  Interventions: Behavioral: Mental Health Treatment
- Telehealth Therapy Treatment: Virtual outpatient therapy
  Interventions: Behavioral: Mental Health Treatment
- No Show Group: Participant who do not attend recommended treatment

INTERVENTIONS:
Behavioral: Mental Health Treatment — Treatment of suicidal ideation
  Groups: Inpatient Treatment; OCIC Treatment; Telehealth Therapy Treatment

SUMMARY:
To address the unmet need of optimizing the treatment and management for adolescent suicidality, the investigators propose to evaluate the effectiveness and safety of telehealth services compared to inpatient and OCIC for suicidal adolescents in target population. To achieve this goal, the investigators propose a multi- site study to compare telehealth, OCIC, and inpatient care, and see which can lead to a lower risk of a suicidal event (primary outcome) as well as higher treatment satisfaction (TS) and satisfaction with life (SL) (secondary outcomes) of both the legal guardians/parents and patients.

DETAILED DESCRIPTION:
The investigators have proposed an observational design. Eligible individuals will be identified during a crisis assessment, either in the emergency department or during an emergency phone or telehealth assessment. Once the individual has been assessed and assigned to the clinician for treatment, study staff will assess if the patient is appropriate for the study using the study eligibility criteria. Individuals who receive treatment in one of the following treatment arms will be eligible for this observation study: inpatient, in-person OCIC or telehealth crisis intervention service. Eligible individuals will be contacted by study staff to introduce and offer the study. If patient and guardian agree, they will complete surveys at baseline and every 2 weeks for 6 months to evaluate outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents that are 12 through 18 years old.
* Adolescents that are brought to the Emergency Department for crisis evaluation due to suicidal thoughts or behaviors.
* Require a higher level of care.
* The presence of a legal guardian for consent.
* Capable of giving signed informed consent/assent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Adolescents with suicidal thoughts who had prior OCIC treatment in the past 12 months.
* Adolescents without the ability to answer survey questions.
* Adolescents that are non-English speaking due to the scales and surveys that are used for this study only being available in English.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescents experiencing suicidal ideation and require a higher level of care.
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Northwell Health, Queens, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No
All data will be de-identified from individual data. Data will only be shared with researchers within the research team.

REFERENCES:
- [Background] Curtin SC, Warner M, Hedegaard H. Increase in Suicide in the United States, 1999-2014. NCHS Data Brief. 2016 Apr;(241):1-8. PMID 27111185
- [Background] QuickStats: Suicide Rates*,dagger for Teens Aged 15-19 Years, by Sex - United States, 1975-2015. MMWR Morb Mortal Wkly Rep. 2017 Aug 4;66(30):816. doi: 10.15585/mmwr.mm6630a6. No abstract available. PMID 28771461
- [Background] Green J, Jacobs B, Beecham J, Dunn G, Kroll L, Tobias C, Briskman J. Inpatient treatment in child and adolescent psychiatry--a prospective study of health gain and costs. J Child Psychol Psychiatry. 2007 Dec;48(12):1259-67. doi: 10.1111/j.1469-7610.2007.01802.x. PMID 18093032
- [Derived] Combs J, Lin PI, DelBello MP, Carle AC, Bridge JA, Axelson DA, Fornari V, Feuer V, Emslie GJ, Kennard BD, Porter SC, Sorter MT, Barzman D. Examining Alternative Treatment Settings for Adolescents With Suicidal Thoughts During the COVID-19 Pandemic. JAACAP Open. 2024 Nov 8;3(3):567-575. doi: 10.1016/j.jaacop.2024.10.005. eCollection 2025 Sep. PMID 40922794

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Inpatient Treatment | OCIC Treatment | Telehealth Therapy Treatment | No Show Group
Started | 87 | 77 | 76 | 9
Completed | 82 | 74 | 74 | 9
Not Completed | 5 | 3 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inpatient Treatment | OCIC Treatment | Telehealth Therapy Treatment | No Show Group | Total
Number analyzed (Participants) | 87 | 77 | 76 | 9 | 249
Age, Continuous [Mean (Full Range); unit: years] | 15.2946 [12.04 to 17.8] | 14.8463 [12.11 to 17.96] | 14.8671 [12.02 to 17.99] | 14.9781 [14.32 to 17.28] | 15.0467 [12.02 to 17.99]
Sex/Gender, Customized [Count of Participants; unit: Participants] — Gender Identity
  Participants
    Male | 20 | 19 | 17 | 2 | 58
    Female | 60 | 46 | 46 | 5 | 157
    Transgender Male (FTM) | 3 | 4 | 5 | 0 | 12
    Transgender Female (MTF) | 0 | 0 | 0 | 0 | 0
    Non-binary | 2 | 5 | 6 | 1 | 14
    Other | 0 | 2 | 0 | 0 | 2
    Choose not to disclose | 2 | 1 | 2 | 1 | 6
Sex: Female, Male [Count of Participants; unit: Participants] — Gender at Birth
  Participants
    Female | 67 | 56 | 58 | 7 | 188
    Male | 20 | 21 | 18 | 2 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 17 | 13 | 2 | 50
  Not Hispanic or Latino | 69 | 60 | 63 | 7 | 199
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 57 | 50 | 51 | 7 | 165
  Black or African American | 10 | 11 | 12 | 0 | 33
  Asian | 1 | 3 | 0 | 0 | 4
  American Indian or Alaskan Native | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Other | 12 | 8 | 5 | 1 | 26
  Mixed Race | 6 | 5 | 8 | 1 | 20
CHRT-SR Score [Mean (Full Range); unit: scores on a scale] — The Concise Health Risk Tracking© Self Report (CHRT-SR), a self-report that focuses on the past week, was designed to assess the severity of current suicide risk. The CHRT-SR assesses both suicidal ideation and other current clinical factors associated with suicide attempts. Scores range from 1 to 56. The higher the overall score represents a worse outcome.
  scores on a scale | 38.0114 [1 to 56] | 32.0657 [1 to 56] | 33.0266 [1 to 56] | 36.7777 [1 to 56] | 34.2634 [1 to 56]

OUTCOME MEASURES:

1. Primary Outcome: Number of Recurrent Suicidal Events Measured by Treatment Arm
Description: Compare the number of recurrent suicidal event across three treatment groups. Suicidal events were measured by hospitalizations during the study time frame in analysis.
Time Frame: 6 Months
Measure: Mean (95% Confidence Interval); unit: hospitalizations
Arm/Group | Inpatient Treatment | OCIC Treatment | Telehealth Therapy Treatment | No Show Group
Number analyzed (Participants) | 87 | 77 | 76 | 9
hospitalizations | 0.66 [0.33 to 0.98] | 0.45 [0.21 to 0.69] | 0.20 [0.08 to 0.31] | 0.60 [-0.08 to 1.28]

2. Secondary Outcome: Which Treatment Leads to Better Life Satisfaction
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Item Bank v1.0 - Short Form 4a was used to measure life satisfaction and response pattern scoring was calculated in RedCap.• Each question has five response options (1 to 5), with the total score ranging from 4 to 20, where higher values indicate better life satisfaction.
Time Frame: 6 Months
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Inpatient Treatment | OCIC Treatment | Telehealth Therapy Treatment | No Show Group
Number analyzed (Participants) | 87 | 77 | 76 | 9
Scores on a scale | 15.75 [13.49 to 18.02] | 16.74 [14.47 to 19.02] | 15.4 [13.33 to 17.48] | 14 [5.83 to 22.16]

3. Other Pre Specified Outcome: Treatment Satisfaction Scores Measured by Treatment Arm
Description: The Client Satisfaction Questionnaire (CSQ), was used to compare the level of treatment satisfaction across three treatment groups. Data collected from children were used in outcome analysis. The four-point Likert scale, with scores from 1 to 4 for each item, provides a total score range of 8 to 32, with higher scores indicating greater satisfaction.
Time Frame: 2 weeks
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Inpatient Treatment | OCIC Treatment | Telehealth Therapy Treatment | No Show Group
Number analyzed (Participants) | 87 | 77 | 76 | 9
Scores on a scale | 23.06 [21.49 to 24.63] | 21.78 [20.34 to 23.21] | 20.9 [19.40 to 22.40] | 17.62 [12.11 to 23.13]

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events were characterized as an increase in suicidal thoughts that resulted in an evaluation in the emergency department, staying overnight in the emergency department, or an emergency visit with a clinician or assessment via phone. Serious adverse events were characterized as an increase in suicidal thoughts that resulted in an inpatient psychiatric hospitalization.
Arm/Group | Inpatient Treatment | OCIC Treatment | Telehealth Therapy Treatment | No Show Group
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/77 | 0/76 | 0/9
Serious Adverse Events (participants affected / at risk) | 20/87 | 13/77 | 12/76 | 3/9
Other Adverse Events (participants affected / at risk) | 12/87 | 9/77 | 13/76 | 3/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inpatient Treatment (N=87) | OCIC Treatment (N=77) | Telehealth Therapy Treatment (N=76) | No Show Group (N=9)
Inpatient psychiatric hospitalization (Psychiatric disorders) | 20 (26) | 13 (15) | 12 (21) | 3 (6) — Participant was admitted to an inpatient psychiatric unit.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inpatient Treatment (N=87) | OCIC Treatment (N=77) | Telehealth Therapy Treatment (N=76) | No Show Group (N=9)
Increase in Suicidal Thoughts Resulting in ED Visit or Other Psychiatric Evaluation (Psychiatric disorders) | 12 (20) | 9 (12) | 13 (15) | 3 (5) — Adverse events were characterized as an increase in suicidal thoughts that resulted in an evaluation in the emergency department, staying overnight in the emergency department, or an emergency visit with a clinician or assessment via phone.

LIMITATIONS AND CAVEATS:
This study is an observational study, which is limited in comparison to an interventional study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT04625686/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT04625686/ICF_001.pdf